CLINICAL TRIAL: NCT01031004
Title: Vistakon Investigational Lens Worn as a Single Use Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-1655
Record Dates: First submitted 2009-11-18; First posted 2009-12-14 (Estimated); Results first posted 2011-03-17 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- narafilcon B (Experimental): contact lens
  Interventions: Device: narafilcon B
- etafilcon A (Active Comparator): contact lens
  Interventions: Device: etafilcon A

INTERVENTIONS:
Device: narafilcon B — contact lens
  Arms: narafilcon B
Device: etafilcon A — contact lens
  Arms: etafilcon A

SUMMARY:
This study is intended to show that the investigational contact lens is clinically equivalent to a currently approved contact lens, when worn as single-use on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* eyes must be best-corrected to a visual acuity of 20/30 or better in each eye
* must be able and willing to wear soft contact lenses on a single use, daily wear basis for the duration of the study
* distance spherical contact lens prescription must be within the range available for the study

Exclusion Criteria:

* systemic diseases which may interfere with contact lens wear
* ocular infection or clinically significant ocular disease
* any previous intraocular surgery
* grade 2 or greater slit lamp findings
* currently pregnant or lactating
* more than 1.00D of refractive astigmatism in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Salt Lake City, Utah
  - Virginia Beach, Virginia
  - Laramie, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Narafilcon B: single use, daily wear contact lens
- Etafilcon A: contact lens worn as single use, daily wear
Period: Overall Study
Arm/Group | Narafilcon B | Etafilcon A
Started | 25 | 25
Completed | 24 | 24
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narafilcon B | Etafilcon A | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (8.19) | 29.2 (8.08) | 29.2 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Findings - Corneal Edema
Description: Investigators examined subjects using a slit lamp and the following scale: 0=none, 1=trace, 2=mild, 3=moderate, 4=severe. This outcome measures the number of eyes that had corneal edema graded 2 or higher at the 1-week visit.
Time Frame: after 1 week of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

2. Primary Outcome: Corneal Edema at Month 1
Description: Number of eyes with corneal edema graded 2 or higher at the 1 month visit. Investigators examined subjects using a slit lamp and the following scale: 0=none, 1=trace, 2=mild, 3=moderate, 4=severe.
Time Frame: after 1 month of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

3. Primary Outcome: Slit Lamp Findings - Corneal Neovascularization
Description: Investigators examined subjects using a slit lamp and the following scale:0=none, 1=trace, 2=mild, 3=moderate, 4= severe. This outcome measures the number of eyes that had corneal neovascularization graded 2 or higher at the 1-week visit.
Time Frame: after 1 week of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

4. Primary Outcome: Slit Lamp Findings - Corneal Neovascularization
Description: as for outcome 3
Time Frame: after 1 month of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

5. Primary Outcome: Slit Lamp Findings - Corneal Staining
Description: Investigators examined subjects using a slit lamp and the following scale:0=none, 1=trace, 2=mild, 3=moderate, 4= severe. This outcome measures the number of eyes that had corneal staining graded 2 or higher at the 1-week visit.
Time Frame: after 1 week of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

6. Primary Outcome: Slit Lamp Findings - Corneal Staining
Description: as for outcome 5
Time Frame: after 1 month of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 1 | 0

7. Primary Outcome: Slit Lamp Findings - Injection
Description: Investigators examined subjects using a slit lamp and the following scale:0=none, 1=trace, 2=mild, 3=moderate, 4= severe. This outcome measures the number of eyes that had injection graded 2 or higher at the 1-week visit.
Time Frame: after 1 week of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

8. Primary Outcome: Slit Lamp Findings - Injection
Description: as for outcome 7
Time Frame: after 1 month of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

9. Primary Outcome: Slit Lamp Findings - Tarsal Abnormalities
Description: Investigators examined subjects using a slit lamp and the following scale:0=none, 1=trace, 2=mild, 3=moderate, 4= severe. This outcome measures the number of eyes that had tarsal abnormalities graded 2 or higher at the 1-week visit.
Time Frame: after 1 week of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

10. Primary Outcome: Slit Lamp Findings - Tarsal Abnormalities
Description: as for outcome 9
Time Frame: after 1 month of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

11. Primary Outcome: Slit Lamp Findings - Infiltrates
Description: Investigators examined subjects using a slit lamp and recorded the presence or absence of infiltrates. This outcome measures the number of eyes that had infiltrates present at the 1-week visit.
Time Frame: after 1 week of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

12. Primary Outcome: Slit Lamp Findings - Infiltrates
Description: as for outcome 11
Time Frame: after 1 month of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0

13. Primary Outcome: Subject Reported Symptoms
Description: Number of eyes in which subjects reported lens-related symptoms after 1 week of lens wear.
Time Frame: after 1 week of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 15 | 8
Statistical Analysis 1: Comparison: Narafilcon B vs Etafilcon A; The hypothesis is that narafilcon B is not statistically different from etafilcon A; Test type: Superiority or Other; p = 0.0466, Fisher Exact

14. Primary Outcome: Subject Reported Symptoms
Description: Number of eyes in which subjects reported lens-related symptoms after 1 month of lens wear.
Time Frame: after 1 month of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 14 | 5
Statistical Analysis 1: Comparison: Narafilcon B vs Etafilcon A; The hypothesis is that narafilcon B is not statistically different from etafilcon A; Test type: Superiority or Other; p = 0.1069, Fisher Exact

15. Primary Outcome: Visual Acuity (VA)
Description: Investigators assessed visual acuity per eye using a Snellen visual acuity chart. This outcome measures the number of eyes, wearing vision correction, that measured visual acuity worse than 20/30 at the 1-week visit.
Time Frame: after 1 week
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0
Statistical Analysis 1: Comparison: Narafilcon B vs Etafilcon A; The hypothesis is that narafilcon B is not statistically different from etafilcon A; Test type: Superiority or Other; p = 0.4605, Chi-squared

16. Primary Outcome: Visual Acuity (VA)
Description: Investigators assessed visual acuity per eye using a Snellen visual acuity chart. This outcome measures the number of eyes, wearing vision correction, that measured visual acuity worse than 20/30 at the 1-month visit.
Time Frame: after 1 month
Population: This analysis includes all participants that completed the study per protocol.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
Number analyzed (eyes) | 48 | 48
eyes | 0 | 0
Statistical Analysis 1: Comparison: Narafilcon B vs Etafilcon A; The hypothesis is that narafilcon B is not statistically different from etafilcon A; Test type: Superiority or Other; p = 0.5774, Chi-squared

17. Primary Outcome: Average Wear Time
Time Frame: after 1 week of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
hours per day | 13.9 (1.91) | 13.7 (2.41)
Statistical Analysis 1: Comparison: Narafilcon B vs Etafilcon A; The hypothesis is that narafilcon B will not be statistically different from etafilcon A; Test type: Superiority or Other; p = 0.6403, t-test, 2 sided

18. Primary Outcome: Average Wear Time
Time Frame: after 1 month of lens wear
Population: This analysis includes all participants that completed the study per protocol.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Narafilcon B | Etafilcon A
Number analyzed (Participants) | 24 | 24
hours per day | 13.6 (2.33) | 13.8 (2.24)
Statistical Analysis 1: Comparison: Narafilcon B vs Etafilcon A; The hypothesis is that narafilcon B is not statistically different from etafilcon A; Test type: Superiority or Other; p = 0.7217, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Narafilcon B | Etafilcon A
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.